CLINICAL TRIAL: NCT05135013
Title: The Association of Hormonal Intake and Demographic Factors With Breast Cancer Risk. An Egyptian Case-controlled Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: NewGiza University (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nermeen Ashoush, Lecturer in Clinical Pharmacy Practice Department, NewGiza University
Other Study IDs: NewGiza University Protocol 1
Record Dates: First submitted 2021-11-16; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Observational Study
Keywords: Hormonal Intake, Breast Cancer Risk, Demographic Factors
MeSH Terms: interventions — Norethindrone Acetate; Ethinyl Estradiol; drospirenone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cases: 1.Cases (100) are those eligible patients who were diagnosed with histopathologically confirmed breast cancer and were during the past 2 years to 2021 (2019-2020).
  Interventions: Drug: Dydrogesterone Tablets, Norethisterone acetate, Ethinyl estradiol, Drospirenone and ethinyl estradiol
- Matched Controls: 2. Matched controls (100) are those participants presenting to the screening clinic and were not diagnosed with breast cancer during the past 2 years to 2021 (2019-2020). Candidates are to be of same range of age (+/-3 years); and similar visiting period (+/-2 months). All controls were confirmed as having no diagnosis of breast cancer, with negative findings on physical breast examination, and breast sono-mammographic screening.
  Interventions: Drug: Dydrogesterone Tablets, Norethisterone acetate, Ethinyl estradiol, Drospirenone and ethinyl estradiol

INTERVENTIONS:
Drug: Dydrogesterone Tablets, Norethisterone acetate, Ethinyl estradiol, Drospirenone and ethinyl estradiol — History of hormonal use as follows:
  1. Reason for hormonal use: contraception, fertility promotion, Polycystic ovary syndrome (PCOS)
  2. Duration of hormonal use
  3. Type of hormonal drug used: dose, hormone type, route of administration

SUMMARY:
The aim of the current study is to investigate the association between hormonal intake, occupational and demographic factors, and the risk of breast cancer (BC) among Egyptian females.

DETAILED DESCRIPTION:
Methodology Design. A case-controlled study.

Setting. Breast cancer clinic and breast cancer screening unit at clinical oncology department, Ain Shams University hospital

Participants.

All cases who will be screened from the BC clinic and the BC screening unit will be assessed for eligibility according to the following inclusion & exclusion criteria:

Inclusion criteria

Age > 18 and < 70

Exclusion criteria

* Diagnosed with other concurrent malignancies.
* A prior history of another cancer.

Eligible candidates will be stratified as cases or matched controls as follows:

1. Cases (100) are those eligible patients who were diagnosed with histopathologically confirmed breast cancer and were during the past 2 years to 2021 (2019-2020).
2. Matched controls (100) are those participants presenting to the screening clinic and were not diagnosed with breast cancer during the past 2 years to 2021 (2019-2020). Candidates are to be of same range of age (+/-3 years); and similar visiting period (+/-2 months). All controls were confirmed as having no diagnosis of breast cancer, with negative findings on physical breast examination, and breast sono-mammographic screening.

Ethical consideration. The protocol will be approved by the ethical committee of NGU and the Clinical Oncology department ASU. The study will be registered at clinicaltrials.gov

Methods.

Data collection for both groups will be done through reviewing of the participants' medical records retrospectively Data collection will include the following data:

* Demographic data: name, age, sex, residence
* Anthropometric data: height, weight, waist & hip circumference & waist to hip ratio and BMI calculation
* Female & menopausal status, age at menarche
* Medical history & comorbidity (CVS, DM 1 or 2, HTN)
* Family history of other cancers, diabetes
* Occupational history
* Social history: smoking, recreational drug use, marital status, nulliparity/multi-parity and lactation
* Dietary habits and diet composition
* Lifestyle habits and degree of regular activity (sedentary, active, etc.)
* History of hormonal use as follows:

  1. Reason for hormonal use: contraception, fertility promotion, PCOS
  2. Duration of hormonal use
  3. Type of hormonal drug used: dose, hormone type, route of administration
* Breast cancer classification:

  1. - Type of pathology - 2- Molecular classification (ER, PR, Her2 receptors status) 3- Staging of BC.

Statistical analysis The frequency distribution of the parameters will be assessed. Parametric data will be presented as mean & standard deviation, while non parametric data will be presented as median & IQR. All data will be analyzed using the appropriate statistical test. Proportions will be presented using number & proportion and will be assessed by the Chi square.

Multiple logistic regression analysis will be used to calculate odds ratios (OR) and corresponding 95% confidence intervals (CI) for the various studied factors in relation to breast cancer occurrence & subtypes.

Moreover, the effect of the combined significant factors to the risk of breast cancer development will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 70

Exclusion Criteria:

* Diagnosed with other concurrent malignancies.
* A prior history of another cancer.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Eligible candidates will be stratified as cases or matched controls as follows:
  1. Cases (100) are those eligible patients who were diagnosed with histopathologically confirmed breast cancer and were during the past 2 years to 2021 (2019-2020).
  2. Matched controls (100) are those participants presenting to the screening clinic and were not diagnosed with breast cancer during the past 2 years to 2021 (2019-2020). Candidates are to be of same range of age (+/-3 years); and similar visiting period (+/-2 months). All controls were confirmed as having no diagnosis of breast cancer, with negative findings on physical breast examination, and breast sono-mammographic screening.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-11-16 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Confirmed Breast Cancer Patients | During the past 2 years to 2021 (2019-2020).
  Patients who were diagnosed with histopathologically confirmed breast cancer and were during the past 2 years to 2021 (2019-2020).

IPD SHARING:
Plan to Share IPD: Undecided